CLINICAL TRIAL: NCT03383900
Title: Inspiratory Muscle Training (EMI) on Inspiratory Muscle Strength, Pulmonary Capacity and Performance in Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grupo de Investigacion en Fisioterapia Cardiovascular y Respiratoria (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Martha Cecilia León Garzón, Doctor en Fisioterapia, Grupo de Investigacion en Fisioterapia Cardiovascular y Respiratoria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PMAFI-12/16
Record Dates: First submitted 2017-11-22; First posted 2017-12-27 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Breathing Exercises: Inspiratory Muscle Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups: experimental (G-IMT) and sham (Gn-IMT). The two groups will perform a protocol of 8 weeks of training (6 days / week) with the PowerBreath
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-IMT (Experimental): The experimental group will first carry out a diaphragmatic reeducation program, followed a posteriori by an inspiratory muscle training program use progressive resistance loads up to 80% of the PImax during the 8 weeks
  Interventions: Device: Inspiratory muscle training
- Gn-IMT (Placebo Comparator): The Gn-IMT will use by an inspiratory muscle training program use resistance loads up to 20% PImax during the 8 weeks.
  Interventions: Device: Inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — The inspiratory muscle training program will be of the "strength and endurance" type, using the POWERbreathe® device and composed of: daily sessions (3 sets of 15 repetitions -inspiration), 6 days a week for 8 weeks. Participants will begin training breathing with a resistance of 20% of their PImax during the first week. After the first week, the resistance will increase between 5% and 10% in each session until reaching 80% of the PImax, which will be maintained during the first month. Upon completion, the PImax value will be re-evaluated and the player will train 80% of this new value during the second month. At the end of the second month, the PImax is evaluated and the player will train the third month with a resistance of 80% of this new value.
  Other Names: G-IMT

SUMMARY:
The training of the respiratory muscles seems to be fundamental in people who require a high physical demand. There is abundant scientific evidence that relates the respiratory variables and the limitation to exercise. The published studies are athletics and cycling, however it is scarce in football. Objective. To assess the effects of inspiratory muscle training on lung function and sports performance in soccer players.

DETAILED DESCRIPTION:
Objective. To assess the effects of inspiratory muscle training (IMT) on lung function, inspiratory muscle strength and athletic performance in soccer players.

Method. Participants will be randomized into two groups: experimental and sham . The two groups will perform a protocol of 8 weeks of training (6 days / week) with the PowerBreathe device. The EG will use progressive resistance loads up to 80% of the MIP, while the SG will use the device with a minimum load (20% PImax) during the 8 weeks. All participants will have the following tests before and after the intervention and 3 months after the end of the program: spirometry (FVC, FEV1), PImax, biophotogrammetry, and fit 30/15 test. For the statistical analysis, a 2-factor variance analysis will be performed for repeated measures and Pearson's correlations. The statistical significance will be set with a value of p <0.05. The effect size will be calculated using the partial eta-square.

ELIGIBILITY:
Inclusion Criteria:

* Soccer players

Exclusion Criteria:

* Soccer players with disabilities

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male soccer players
Enrollment: 22 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
RESPIRATORY CAPACITY | 1 week
  The variable PImax. will be measured through spirometry whose value will be expressed in cm / H2O

SECONDARY OUTCOMES:
Biofotogrametry | 1 week
  Biofotogrametry is a tool used to measure the thoracic expansion, the respiratory pattern and its cadence; by recording a video of the breathing pattern that observes the pre- and post-breathing of the subjects.
  The unit of measurement in which the results are expressed for the variable thoracic extension will be in cm, and for the respiratory pattern and its percentage cadence (%).
Sports performance | 1 week
  The performance variable will be evaluated using the "fit" 30/15 test, a tool used in athletes to determine the maximum intermittent aerobic speed (VO2max); the results of this test allow later to plan the specific training protocol of the sports team.
Lactate in blood | 1 week
  The amount of blood lactate will be measured after inspiratory muscle training with a lactate meter, its results will be expressed in the unit of measure mg / dL.
Static equilibrium | 1 week
  Static equilibrium was obtained through an analysis of stabilometric variables on an equilibrium platform. The players had to stand on the platform with bipodal support (45º) for 90 seconds with eyes open and 90 seconds with eyes closed. During the measurement with their eyes open, the players had to keep their gaze on a fixed point that coincided with the height of their eyes and was about 2.5 meters from the platform. A FreeStep platform (Rome, Italy) was used

CONTACTS AND LOCATIONS:
Overall Officials: Martha C León Garzón, Therapy, Principal Investigator — Catholic university San Antonio of Murcia
Locations (2):
- Spain (2):
  - Catholic University San Antonio of Murcia, Murcia
  - Mayayo Sports Center, Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozmen T, Gunes GY, Ucar I, Dogan H, Gafuroglu TU. Effect of respiratory muscle training on pulmonary function and aerobic endurance in soccer players. J Sports Med Phys Fitness. 2017 May;57(5):507-513. doi: 10.23736/S0022-4707.16.06283-6. Epub 2016 Feb 12. PMID 28399624
- [Background] Guy JH, Edwards AM, Deakin GB. Inspiratory muscle training improves exercise tolerance in recreational soccer players without concomitant gain in soccer-specific fitness. J Strength Cond Res. 2014 Feb;28(2):483-91. doi: 10.1519/JSC.0b013e31829d24b0. PMID 23722111
- [Background] Nicks CR, Morgan DW, Fuller DK, Caputo JL. The influence of respiratory muscle training upon intermittent exercise performance. Int J Sports Med. 2009 Jan;30(1):16-21. doi: 10.1055/s-2008-1038794. Epub 2008 Oct 30. PMID 18975258